CLINICAL TRIAL: NCT06017336
Title: Investigation of the Effects of Inspiratory Muscle Training on Oxygen Consumption, Muscle Oxygen and Physical Activity Level in Patients With Parkinson's Disease
Brief Title: Effects of Inspiratory Muscle Training in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Cardiopulmonary Physiotherapy and Rehabilitation, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gazi University 78
Record Dates: First submitted 2023-08-15; First posted 2023-08-30 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; inspiratory muscle training; oxygen consumption; physical activity
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Control Groups; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training Group (Experimental): Patients in the training group will be performed inspiratory muscle training with the PowerBreathe® (inspiratory muscle training device) device at 50% of the maximal inspiratory pressure.
  Interventions: Other: Inspiratory Muscle Training Group
- Control Group (Sham Comparator): Control group will be given breathing exercises as a home program for 8 weeks.
  Interventions: Other: Control Group (breathing exercises)

INTERVENTIONS:
Other: Inspiratory Muscle Training Group — Patients in the inspiratory muscle training group will be given inspiratory muscle strength training with the Powerbreathe® (inspiratory muscle training device) device at 50% of the maximal inspiratory pressure, 2 sets of 15 minutes a day for a total of 30 min/day or a single set of 30 min/day, 7 days/week for 8 weeks. Patients in the inspiratory muscle training group will continue their respiratory muscle strength training with a home program 6 days a week under the supervision of a physiotherapist 1 day a week. The MIPs of the patients will be re-measured every week and the training workload will be determined at 50% of the new maximal inspiratory pressure.
  Arms: Inspiratory Muscle Training Group
Other: Control Group (breathing exercises) — Thoracic expansion exercises will be given to the control group as a home program. The control group will be asked to do thoracic expansion exercises seven days/week and 120 times/day for eight weeks. The patients in the control group will be called once a week to check their home schedules, and they will be asked to keep a diary.
  Arms: Control Group

SUMMARY:
Parkinson's patients usually have a significant decrease in respiratory muscle strength and respiratory function, which may increase in proportion to the severity of the disease. In addition, peripheral muscles may become dysfunctional by the rigidity caused by the disease. This reduces exercise capacity and may lead to a decrease in oxygen consumption. Respiratory muscle training has increased respiratory muscle strength in people with Parkinson's Disease (PD). However, its effectiveness on other functional outcomes has not been determined and studied.

DETAILED DESCRIPTION:
Parkinson's disease is the second most common neurodegenerative disease. The main motor symptoms seen in Parkinson's disease are tremors, rigidity, bradykinesia, and decreased postural reflexes. In addition, respiratory problems that lead to death may often be seen. This is caused by dysfunction in the respiratory muscles and postural abnormalities, as well as changes in upper airway muscle activation and coordination. The coughing or exhaling reflex requires coordinated motor activity, and inadequate airway defence puts patients at risk for pneumonia. Aspiration into the lower airways results in a distinct series of events, including coughing and swallowing as the first attempt to clear the airway. Aspiration pneumonia is seen in Parkinson's patients because the coordination of these processes is unsuccessful, and the cough force is insufficient. Upper airway obstruction may occur due to stiffness and fatigue in the thyroarytenoid muscles. In addition, pathological processes such as bradykinesia, coordination disorder, and inspiratory muscle weakness can cause kyphoscoliosis and a decrease in lung volumes, resulting in restrictive respiratory function abnormality due to decreased chest wall compliance due to rigidity. In Parkinson's disease, respiratory muscles, like other skeletal muscles, are affected by stiffness, and weakness of the respiratory muscles makes it difficult to overcome this stiffness, resulting in reduced lung volumes. It is thought that this condition may develop due to the decrease in elastic retraction of the chest wall. In addition, mitochondrial dysfunction due to the pathogenesis of the disease also leads to deterioration in muscle oxygen metabolism. In individuals with reduced muscle oxygen, exercise tolerance and muscle strength decrease. Autonomic dysfunction of varying severity is observed in almost all patients, depending on the degeneration of spinal autonomic neurons or the side effects of dopaminergic that are part of pharmacological treatment. Patients may experience increased fatigue as well as autonomic dysfunction. Inadequate oxygen delivery and utilization to the muscles may limit skeletal muscle oxygenation and lead to increased use of anaerobic systems, resulting in fatigue. This causes a decrease in the level of physical activity and reduces the quality of life.

However, studies investigating the effects of inspiratory muscle training in Parkinson's patients are insufficient. The aim of this study is to investigate the effects of inspiratory muscle training on maximum and functional exercise capacity, muscle oxygen, peripheral and respiratory muscle strength, respiratory muscle endurance, respiratory function, dyspnea, fatigue, cough strength, autonomic dysfunction, physical activity level and quality of life in patients with Parkinson's disease.For this purpose, our study was planned as a randomized, controlled, three-blind (investigators, patient, and analyzer) prospective study. According to the block randomization result, at least 20 patients with a diagnosis of Parkinson's Disease will be included in the training and control groups.

Patients in the inspiratory muscle training group will be given inspiratory muscle strength training with the Powerbreathe device at 50% of the maximal inspiratory pressure for a total of 8 weeks, for a total of 30 minutes a day. Thoracic expansion exercises will be given to the control group as a home program for 8 weeks. All assessments will be completed in two days, before and after eight weeks of training.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 45-80,
2. Follow-up with a diagnosis of Parkinson's disease for more than six months
3. Stages I-III according to the modified Hoehn and Yahr scale
4. Parkinson's patients with independent walking capacity will be included.

Exclusion Criteria:

1. Having a neurological disease other than Parkinson's disease
2. Patients with a diagnosed lung disease that may affect respiratory functions
3. At least 10 pack years or more of smoking history
4. According to the American Association of Sports Medicine (ACSM) with absolute and relative contraindications to exercise tests
5. Those with a Mini-Mental State Rating Scale score of less than 18
6. Patients with additional cardiac orthopaedic and psychological problems that limit the evaluation will be excluded from the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Oxygen Consumption | Trough study completion, an average of 2 year
  Cardiopulmonary Exercises Test

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Trough study completion, an average of 2 year
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were
Respiratory Muscle Endurance | Trough study completion, an average of 2 year
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load.
Pulmonary function (Forced vital capacity (FVC) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced vital capacity (FVC) will be measured.
Pulmonary function (Forced expiratory volume in the first second (FEV1) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced expiratory volume in the first second (FEV1) will be measured.
Pulmonary function (FEV1 / FVC) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. FEV1 / FVC will be measured.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be measured.
Pulmonary function (Peak flow rate (PEF)) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Peak flow rate (PEF) will be measured.
Peripheral Muscle Strength | Trough study completion, an average of 2 year
  Peripheral muscle strength will be evaluated with a dynamometer.
Lower extremity exercise capacity | Trough study completion, an average of 2 year
  Lower extremity exercise capacity will be evaluated with six- minute walking test.
Upper extremity exercise capacity | Trough study completion, an average of 2 year
  Upper extremity exercise capacity will be evaluated with the six-minute pegboard and ring test (6-PBRT).
Cough Strength | Trough study completion, an average of 2 year
  Cough strength will be assessed using a peak cough flow meter (PEFmeter) (ExpiRite Peak Flow Meter, China).
Autonomic dysfunction | Trough study completion, an average of 2 year
  It will be measured by postural change during ECG recording
Fatigue Severity | Trough study completion, an average of 2 year
  Fatigue will be evaluated using the Parkinson Fatigue Scale. Total score varies between 16-80. As the score increases, the severity of fatigue increases.
Life quality | Trough study completion, an average of 2 year
  Patients' health-related quality of life will be evaluated using the Parkinson's disease questionnaire-39. The total score varies between 0-156, and the quality of life worsens as the score increases.
Muscle oxygenation | Trough study completion, an average of 2 year
  Muscle oxygenation assessment will be performed using the Moxy monitor (Moxy, Fortiori Design LLC, Minnesota, USA).
Physical Activity Level | Trough study completion, an average of 2 year
  A multi-sensor activity monitor will be used to assess the level of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Musa GÜNEŞ, MsC, Principal Investigator — Gazi University; Hatice Ayşe TOKÇAER BORA, Prof. Dr., Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reyes A, Castillo A, Castillo J, Cornejo I. The effects of respiratory muscle training on peak cough flow in patients with Parkinson's disease: a randomized controlled study. Clin Rehabil. 2018 Oct;32(10):1317-1327. doi: 10.1177/0269215518774832. Epub 2018 May 13. PMID 29756459
- [Background] Reyes A, Castillo A, Castillo J, Cornejo I, Cruickshank T. The Effects of Respiratory Muscle Training on Phonatory Measures in Individuals with Parkinson's Disease. J Voice. 2020 Nov;34(6):894-902. doi: 10.1016/j.jvoice.2019.05.001. Epub 2019 May 31. PMID 31155431
- [Background] McMahon L, Blake C, Lennon O. Nonpharmacological interventions for respiratory health in Parkinson's disease: A systematic review and meta-analysis. Eur J Neurol. 2021 Mar;28(3):1022-1040. doi: 10.1111/ene.14605. Epub 2020 Dec 1. PMID 33098349
- [Background] Mohammed Yusuf SF, Bhise A, Nuhmani S, Alghadir AH, Khan M. Effects of an incentive spirometer versus a threshold inspiratory muscle trainer on lung functions in Parkinson's disease patients: a randomized trial. Sci Rep. 2023 Feb 13;13(1):2516. doi: 10.1038/s41598-023-29534-8. PMID 36781936
- [Background] Huang CC, Lai YR, Wu FA, Kuo NY, Cheng BC, Tsai NW, Kung CT, Chiang YF, Lu CH. Detraining Effect on Pulmonary and Cardiovascular Autonomic Function and Functional Outcomes in Patients With Parkinson's Disease After Respiratory Muscle Training: An 18-Month Follow-Up Study. Front Neurol. 2021 Oct 21;12:735847. doi: 10.3389/fneur.2021.735847. eCollection 2021. PMID 34744975
- [Derived] Gunes M, Bosnak Guclu M, Guvenir A, Bora Tokcaer A. Effects of inspiratory muscle training on upper and lower extremity functional exercise capacity, muscle oxygen, and cough strength in patients with Parkinson's disease. Physiother Theory Pract. 2025 Dec 14:1-14. doi: 10.1080/09593985.2025.2602854. Online ahead of print. PMID 41392483